CLINICAL TRIAL: NCT00868296
Title: A Muliticenter, Open Label Safety Study of 2 Doses of Pantoprazole Sodium Enteric-Coated Spheroid Suspension in Infants Aged Less Than 12 Months With Presumed GERD
Brief Title: Open Label Safety Study of Enteric-Coated Spheroid Suspension in Infants Aged Less Than 12 Months With Presumed Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3001B3-335
Record Dates: First submitted 2009-03-20; First posted 2009-03-24 (Estimated); Results first posted 2010-01-07 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-04

CONDITIONS: Gastroesophageal Reflux
Keywords: Safety
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

ARMS (2):
- Low dose (Active Comparator)
  Interventions: Drug: pantoprazole
- High dose (Active Comparator)
  Interventions: Drug: pantoprazole

INTERVENTIONS:
Drug: pantoprazole

SUMMARY:
The purpose of this study is to provide additional information on safety and tolerability after multiple does of pantoprazole. Only patients who successfully completed the 3001B3-331 study (NCT00362609) or 3001B3-333 study (NCT00259012) are eligible to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of the 3001B3-331 study (NCT00362609) or 3001B3-333 study (NCT00259012) Study.

Exclusion Criteria:

* Patients requiring chronic use of warfarin, carbamepazine, or phenytoin.

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For Germany, medinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For South Africa, ZAFinfo@wyeth.com; Trial Manager, Principal Investigator — For Australia, medinfo@wyeth.com; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com; Trial Manager, Principal Investigator — For Italy, descresg@wyeth.com; Trial Manager, Principal Investigator — For Switzerland, med@wyeth.com
Locations (70):
- United States (45):
  - Phoenix, Arizona
  - Loma Linda, California
  - Oakland, California
  - Orange, California
  - Sacramento, California
  - San Diego, California
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Miami, Florida
  - Sunrise, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Lexington, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Flint, Michigan
  - Omaha, Nebraska
  - Camden, New Jersey
  - New Brunswick, New Jersey
  - Newark, New Jersey
  - Albany, New York
  - Brooklyn, New York
  - New York, New York
  - The Bronx, New York
  - Valhalla, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Danville, Pennsylvania
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Richmond, Virginia
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Brisbane, Australia
- Belgium (2):
  - Edegem
  - Leuven
- Canada (5):
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec
- Paris, France
- Germany (3):
  - Bochum
  - Osnabrück
  - Potsdam
- Italy (3):
  - Brescia
  - Napoli
  - Roma
- Rotterdam, Netherlands
- Poland (3):
  - Bydgoszcz
  - Krakow
  - Lublin
- South Africa (5):
  - Panorama, CPT
  - Pietermaritzburg, KwaZulu-Natal
  - Durban
  - Overport
  - Pretoria
- Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited worldwide March 2006 to February 2008.
Pre-assignment Details: Patients were eligible for enrollment into the study after completion of either study 3001B3-331 (NCT00362609) or study 3001B3-333 (NCT00259012).
Groups:
- Low Dose Pantoprazole: Patients who participated previously in study 3001B3-333 (NCT00259012) (infants) and weighed 2.5 to <7 kg generally received pantoprazole sodium enteric-coated spheroid suspension daily 2.5 mg; those weighing ≥ 7 kg to ≤ 15 kg generally received pantoprazole sodium enteric-coated spheroid suspension daily 5 mg. (A patient's dose may have been increased from the dose used in the previous study at the start of this open label extension study to manage clinical symptoms) No patients who participated previously in study 3001B3-331 (NCT00362609) (pre-term/neonates) were included in the low dose group.
- High Dose Pantoprazole: Patients who participated previously in study 3001B3-333 (NCT00259012) (infants) and weighed 2.5 to <7kg generally received pantoprazole sodium enteric-coated spheroid suspension daily 5 mg; those weighing ≥ 7 kg to ≤ 15 kg generally received pantoprazole sodium enteric-coated spheroid suspension daily 10 mg. (A patient's dose may have been increased from the dose used in the previous study at the start of this open label extension study to manage clinical symptoms.) All patients who participated previously in study 3001B3-331 (NCT00362609) (pre-term/neonates) received 2.5 mg (or higher, if the dose was increased at the start of this open label extension study to manage clinical symptoms) and were classified as part of the high dose group for analysis purposes.
Period: Overall Study
Arm/Group | Low Dose Pantoprazole | High Dose Pantoprazole
Started | 12 | 46
Completed | 12 | 43
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Pantoprazole | High Dose Pantoprazole | Total
Number analyzed (Participants) | 12 | 46 | 58
Age Continuous [Mean (Standard Deviation); unit: months] | 7.34 (3.06) | 5.55 (3.44) | 5.92 (3.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 21 | 26
  Male | 7 | 25 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Laboratory Test Values of Potential Clinical Importance During Treatment Period
Description: Pre-defined criteria were established for each laboratory test to define the values that would be identified as of potential clinical importance. Criteria are as follows: Potassium ≤ 3.0 mEq/L or ≥ 6.2 mEq/L; Carbon dioxide < 12 mEq/L or > 35 mEq/L; Total bilirubin > 1.5xULN; CPK > 3xULN; Gastrin ≥ 600 pg/mL; Neutrophils < 10% or > 80%; Platelet count < 100 x10 to the third power/ul or > 600 x10 to the third power/ul; Urine protein albumin > 2+ (dipstick) 100mg/dL or positive; Urine leukocyte esterase > 2+ (dipstick) moderate or positive.
Time Frame: 6 weeks
Population: Patients who received ≥1 dose of pantoprazole and had laboratory test results. The number of patients (n) tested varied by test, variations shown (low dose, high dose): Carbon dioxide (n=7,26), CPK (n=12,42), Gastrin (n=9,25), Neutrophils (n=12,44), Platelet count (n=12,41), Urine protein albumin (n=10,38), Urine leukocyte esterase (n=10,38).
Measure: Number; unit: patients
Arm/Group | Low Dose Pantoprazole | High Dose Pantoprazole
Number analyzed (Participants) | 12 | 45
patients
  Potassium (mmol/L) | 0 | 3
  Carbon dioxide (mmol/L) | 0 | 1
  Total bilirubin (µmol/L) | 0 | 1
  CPK (mU/mL) | 0 | 2
  Gastrin (pg/mL) | 0 | 1
  Neutrophils (1,000,000,000/L) | 1 | 0
  Platelet count (1,000,000,000/L) | 0 | 2
  Urine protein albumin | 0 | 1
  Urine leukocyte esterase | 1 | 3

2. Primary Outcome: Growth Parameters Z-scores
Description: Z-Score is a statistical measure to evaluate how a single data point compares to a standard. A Z-Score describes whether a mean is above or below the standard and how unusual the measurement is. Z-scores primarily range from -3 to +3. A Z-score of 0 indicates the same mean, >0 a greater mean, and <0 a lesser mean than the standard. In this study, infant growth parameters were compared to a standard defined by Centers for Disease Control's growth charts.
Time Frame: 6 weeks
Population: Safety population (all patients with ≥1 dose of study drug) who also had baseline and end of study evaluations. Data point pairs were analyzed. All patients in study 3001B3-335 originated from study 3001B3-331 or -333 and baselines from the original study they were in were used.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Low Dose Pantoprazole | High Dose Pantoprazole
Number analyzed (Participants) | 12 | 46
units on scale
  Length - Baseline (n=12, 45) | 0.33 (1.11) | -1.63 (2.99)
  Length - Final evaluation (n=12, 45) | 0.45 (1.29) | -1.04 (2.52)
  Weight - Baseline (n=12, 46) | -0.16 (1.15) | -1.26 (1.90)
  Weight - Final evaluation (n=12, 46) | -0.05 (1.33) | -1.00 (1.73)
  Head circumference - Baseline (n=11, 45) | 0.31 (1.17) | -1.06 (2.10)
  Head circumference - Final evaluation (n=11, 45) | 0.25 (1.21) | -0.62 (1.71)
Statistical Analysis 1: Comparison: Low Dose Pantoprazole vs High Dose Pantoprazole; Between group comparison for change from baseline in length z-score; Test type: Superiority or Other; p = 0.857, ANCOVA — Analysis with treatment as factor; baseline as covariate
Statistical Analysis 2: Comparison: Low Dose Pantoprazole vs High Dose Pantoprazole; Between group comparison for change from baseline in weight z-score; Test type: Superiority or Other; p = 0.901, ANCOVA — Analysis with treatment as factor; baseline as covariate
Statistical Analysis 3: Comparison: Low Dose Pantoprazole vs High Dose Pantoprazole; Between group comparison for change from baseline in head circumference z-score; Test type: Superiority or Other; p = 0.807, ANCOVA — Analysis with treatment as factor; baseline as covariate
Statistical Analysis 4: Comparison: Low Dose Pantoprazole; Final evaluation compared to baseline within group comparison for length z-score; Test type: Superiority or Other; p = 0.595, t-test, 2 sided; paired
Statistical Analysis 5: Comparison: High Dose Pantoprazole; Final evaluation compared to baseline within group comparison for length z-score; Test type: Superiority or Other; p = 0.016, t-test, 2 sided; paired
Statistical Analysis 6: Comparison: Low Dose Pantoprazole; Final evaluation compared to baseline within group comparison for weight z-score; Test type: Superiority or Other; p = 0.347, t-test, 2 sided; paired
Statistical Analysis 7: Comparison: High Dose Pantoprazole; Final evaluation compared to baseline within group comparison for weight z-score; Test type: Superiority or Other; p = 0.040, t-test, 2 sided; paired
Statistical Analysis 8: Comparison: Low Dose Pantoprazole; Final evaluation compared to baseline within group comparison for head circumference z-score; Test type: Superiority or Other; p = 0.892, t-test, 2 sided; paired
Statistical Analysis 9: Comparison: High Dose Pantoprazole; Final evaluation compared to baseline within group comparison for head circumference z-score; Test type: Superiority or Other; p = 0.006, t-test, 2 sided; paired

ADVERSE EVENTS:
Arm/Group | Low Dose Pantoprazole | High Dose Pantoprazole
Serious Adverse Events (participants affected / at risk) | 1 | 2
Other Adverse Events (participants affected / at risk) | 8 | 30
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Low Dose Pantoprazole | High Dose Pantoprazole
Gastroenteritis (Gastrointestinal disorders) | 1/12 | 0/46
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0/12 | 1/46
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/12 | 1/46
Otitis media (Ear and labyrinth disorders) | 1/12 | 0/46
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Low Dose Pantoprazole | High Dose Pantoprazole
Accidental injury (General disorders) | 0/12 | 1/46
Fever (General disorders) | 1/12 | 4/46
Hernia (General disorders) | 0/12 | 1/46
Immune system disorder (General disorders) | 1/12 | 0/46
Infection (General disorders) | 1/12 | 0/46
Injection site pain (General disorders) | 0/12 | 1/46
Bradycardia (Cardiac disorders) | 0/12 | 1/46
Tachycardia (Cardiac disorders) | 0/12 | 1/46
Constipation (Gastrointestinal disorders) | 0/12 | 3/46
Diarrhea (Gastrointestinal disorders) | 0/12 | 1/46
Gastroenteritis (Gastrointestinal disorders) | 0/12 | 2/46
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2/12 | 1/46
Gingivitis (Gastrointestinal disorders) | 0/12 | 1/46
Mouth ulceration (Gastrointestinal disorders) | 0/12 | 1/46
Oral moniliasis (Gastrointestinal disorders) | 0/12 | 1/46
Tooth disorder (Gastrointestinal disorders) | 1/12 | 4/46
Vomiting (Gastrointestinal disorders) | 1/12 | 3/46
Ecchymosis (Blood and lymphatic system disorders) | 0/12 | 1/46
Creatine phosphokinase increased (Metabolism and nutrition disorders) | 0/12 | 1/46
Healing abnormal (Metabolism and nutrition disorders) | 0/12 | 1/46
Hypophosphatemia (Metabolism and nutrition disorders) | 0/12 | 1/46
Musculoskeletal anomaly (Musculoskeletal and connective tissue disorders) | 0/12 | 1/46
Agitation (Nervous system disorders) | 0/12 | 1/46
Hostility (Nervous system disorders) | 0/12 | 1/46
Insomnia (Nervous system disorders) | 1/12 | 0/46
Apnea (Respiratory, thoracic and mediastinal disorders) | 0/12 | 1/46
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0/12 | 1/46
Cough increased (Respiratory, thoracic and mediastinal disorders) | 2/12 | 3/46
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0/12 | 1/46
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1/12 | 1/46
Pulmonary physical finding (Respiratory, thoracic and mediastinal disorders) | 1/12 | 0/46
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0/12 | 1/46
Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0/12 | 1/46
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/12 | 1/46
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 4/12 | 4/46
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0/12 | 1/46
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2/12 | 3/46
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0/12 | 1/46
Eczema (Skin and subcutaneous tissue disorders) | 0/12 | 3/46
Erythema (Skin and subcutaneous tissue disorders) | 1/12 | 0/46
Herpes simplex (Skin and subcutaneous tissue disorders) | 0/12 | 1/46
Maculopapular rash (Skin and subcutaneous tissue disorders) | 0/12 | 1/46
Pustular rash (Skin and subcutaneous tissue disorders) | 1/12 | 0/46
Rash (Skin and subcutaneous tissue disorders) | 1/12 | 2/46
Blepharitis (Eye disorders) | 0/12 | 1/46
Conjunctivitis (Eye disorders) | 0/12 | 2/46
Ear pain (Ear and labyrinth disorders) | 0/12 | 1/46
Eye disorder (Eye disorders) | 1/12 | 0/46
Otitis media (Ear and labyrinth disorders) | 2/12 | 5/46
Vaginal moniliasis (Reproductive system and breast disorders) | 0/12 | 1/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.